CLINICAL TRIAL: NCT05151172
Title: A Multicentre, Prospective, Randomized, Parallel Group, Open-label Design to Determine the Efficacy and Safety of Endovascular Thrombectomy for Ischemic Stroke Patients With Symptomatic Acute Medium Vessel Intracranial Occlusions
Brief Title: EndovaSCular TreAtment to imProve outcomEs for Medium Vessel Occlusions (ESCAPE-MeVO Trial)
Acronym: ESCAPE-MeVO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Michael D Hill (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor-Investigator, Dr. Michael D Hill, Professor, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version E, November 15, 2023
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Acute Ischemic Stroke
Keywords: endovascular thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: ESCAPE-MeVO is a multicenter, prospective, randomized, open- label study with blinded endpoint evaluation (PROBE design). Subjects will be allocated (1:1) to best guideline-based best medical care plus endovascular therapy (EVT) vs. best guideline- based best medical care alone.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- best medical care (Placebo Comparator): All patients will receive the best standard of medical care according to modern acute stroke care guidelines All patients including the ones in control arm will receive the best standard of medical care according to modern acute stroke care guidelines. The model will be the Canadian best practices guidelines for acute stroke care. These are very similar to the guidelines of the American Stroke Association and the European Stroke Organization. All participants are expected to be admitted to hospital as part of routine standard of care.It is expected that all participants will undergo a routine work-up for the mechanism of their stroke and be treated appropriately and definitively.
  Interventions: Other: Standarad medical care
- endovascular thrombectomy (Experimental): All participants will receive the best standard of medical care according to modern acute stroke care guidelines. In the intervention/experimental arm, participants will be treated with endovascular thrombectomy with a Solitaire device (Medtronic) as the first line approach. The trial mandates that the first attempt is performed with a Solitaire X device (3mm, 4mm or 6mm diameter devices; Medtronic). The remaining treatment technique is left to the discretion of the treating neurointerventionalist. Secondary devices may be used if success is not achieved after use of the first device.
  Interventions: Device: endovascular thrombectomy (EVT)

INTERVENTIONS:
Device: endovascular thrombectomy (EVT) — minimally invasive endovascular surgery for mechanical removal of occluding intracranial thrombus
  Other Names: solitaire X
  Arms: endovascular thrombectomy
Other: Standarad medical care — Stanadard medical care wil involve use of thrombolytic drugs, Blood pressure management, use of antiplatelet or anti coagulant drugs
  Arms: best medical care

SUMMARY:
Stroke occurs when a blood clot causes a blockage in a blood vessel (artery) within the brain. This type of stroke is called an ischemic stroke and carries a high risk of disability or death. Stroke must be treated very fast. Any delay of even 10 minutes can result in the difference between an independent and a disabled outcome, and in some cases between life and death. Endovascular therapy (EVT) or Thrombectomy is a procedure to remove the blood clot (thrombus) from a blood vessel to reopen it (recanalization). Patients are likely to benefit from a thrombectomy procedure when it is performed in a larger blood vessel. Currently it is not known if thrombectomy procedure will benefit the patients presenting with the stroke that has been caused by a blood clot in a medium sized blood vessel (medium vessel occlusion, MeVO). This trial will enrol patients diagnosed with acute stroke due to a clot in the medium sized vessel. The patients will be randomized within 12 hours of their symptom onset to either standard of care or standard of care plus thrombectomy procedure. The participation will last for 12 months Escape MeVO coordinating centre is located at the University of Calgary. There will be up to 75 sites. We will be recruiting a total of 530 patients.

DETAILED DESCRIPTION:
ESCAPE-MeVO is a multicenter, prospective, randomized, open- label study with blinded endpoint evaluation (PROBE design). Participants will be randomized to routine best medical stroke care governed by current guidelines (control group) or to EVT plus best medical care. EVT will be performed with one of the Solitaire group of intracranial stent-retriever devices (Solitaire X, Medtronic) as the first line approach according to the manufacturers' specifications for use.

Patients with clinical symptoms of acute stroke, last seen normal within the last 12 hours, and with either NIHSS ≥ 5 or NIHSS 3-5 due to disabling symptoms in the judgement of the stroke team shall undergo imaging to identify the MeVO and assess the status of the affected brain parenchyma. As is being currently practiced across different stroke centers, imaging may follow different imaging paradigms:

* Option 1: NCCT + mCTA (first phase covers intracranial and extracranial vessels)
* Option 2: NCCT + mCTA/spCTA + either mCTA tissue level perfusion maps or CTP perfusion maps
* Option 3: DWI-MRI + MRA (of both the intracranial and extracranial vessels). Approach to the EVT procedure and technique will be at the discretion of the interventionist and team, with the exception that the first thrombectomy attempt is performed with one of the Solitaire group of intracranial stent-retriever devices (Solitaire X, Medtronic). Available, approved off-the-shelf, secondary devices may be used if reperfusion success is not achieved after use of the first device, at the discretion of the neuro-interventionalist

This study consists of one 90-day study period for each participant. Participants will be hospitalized for care after their acute stroke according to the current standard of care. Participants are required to return to clinic on Day 90 for end-of-study assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke clinically eligible for immediate EVT
2. Age ≥18 years at the date of randomization
3. Time from onset (or last-seen-well) to randomization <12 hours
4. Disabling stroke defined as follows:

   1. baseline National Institutes of Health Stroke Scale (NIHSS) score >5 at the time of randomization
   2. NIHSS 3-5 with disabling deficit (eg. hemianopia, aphasia, loss of hand function) as determined by the attending physician in context of the patient's life situation
5. Confirmed symptomatic and endovascularly treatable MeVO based on neurovascular non-invasive imaging (mCTA or MRA), at one or more of the following locations: M2 or M3 segment, A2 or A3 segment, P2 or P3 segment1.
6. . Clinical deficit commensurate with MeVO occlusion location
7. . Signed informed consent, two-physician consent, or deferral of consent where approved

   Exclusion Criteria:
8. ASPECTS ≤ 5
9. The following depend on the imaging modality of the participating site:

9a. NCCT + mCTA

* Well demarcated hypodensity in the majority of the brain parenchyma supplied by the occluded vessel or absence of collaterals in the affected territory on the delayed phases of the mCTA OR 9b. NCCT + (m)CTA + CTP**
* Lack of core: penumbra mismatch (if the CTP is uninterpretable, e.g., due to motion artifacts, apply exclusion criteria from 9a. If single-phase CTA is performed, score collaterals accordingly. If NCCT + mCTA + CTP are all performed, the core: penumbra mismatch criteria are sufficient for exclusion) OR 9c. MRI
* Diffusion restriction in the majority of the brain parenchyma supplied by the occluded vessel
* if MR perfusion is performed: lack of core:penumbra mismatch 10) Any evidence of intracranial hemorrhage on qualifying imaging 11) Patients living in a nursing home or requiring daily nursing care or assistance with activities of daily living.

  12) Patient has a major co-morbid illness, such as severe dementia, advanced cancer, advanced heart failure etc. such that they are unlikely to be able to complete follow-up or they are unlikely to achieve the primary outcome due to the underlying illness (rather than the stroke or its treatment).

  13) Pregnancy: female with positive urine or serum beta human chorionic gonadotropin (β-hCG) test 14) Participation in another clinical therapeutic intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale score (mRS) | 90 days after randomization
  global neurological functional outcome measured on the modified Rankin Scale

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 24 Hour
  Stroke scale
Mortality | 90 days
  All cause mortality
European Quality of LIfe Scale (EQ-5D-5L) | 90 days
  Self reported health status

CONTACTS AND LOCATIONS:
Overall Officials: Mayank Goyal, MD, Principal Investigator — University of Calgary and Foothills Medical Centre
Locations (53):
- United States (20):
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Sutter Health, San Francisco, California
  - Providence Little company of Mary, Torrance, California
  - Yale School of Medicine, New Haven, Connecticut
  - Baptist Health Medical Centre, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northwestern Medicine, Chicago, Illinois
  - Rush university Medical Centre, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - bBston Medican Center, Boston, Massachusetts
  - Mount Sinai Health System, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Ohio Health (Columbus ORI), Columbus, Ohio
  - University of Toledo, Toledo, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of TN Health Sciences Centre, Memphis, Tennessee
  - Texas stroke Institute, Plano, Texas
  - Swedish Medical Centre, Seattle, Washington
- Canada (14):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver general hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II HSC, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton Health sciences, Hamilton, Ontario
  - London Health Sciences, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Germany (6):
  - Klinikum Altenburger Lang, Altenburg
  - Albert-Ludwigs-Universität Freiburg, Freiberg
  - University of Heidelberg, Heidelberg
  - University Hospital Tübingen, Tübingen
  - University Hospital of Bonn, Venusberg
  - Wurzberg University Hospital, Würzburg
- United Kingdom (13):
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Royal Victoria Hospital, Belfast
  - Cambridge University Hospital, Cambridge
  - Hull University Teaching Hospital, Hull
  - Leeds Teaching Hospitals, Leeds
  - The Royal London Hospital, London
  - Kings college Hospital, London
  - St Georges Hospital, London
  - Charing Cross Hospital, London
  - University College London Hospital, London
  - Nottingham University Hospital, Nottingham
  - John Radcliffe Hopital, Oxford
  - University Hospital Southhampton, Southampton

IPD SHARING:
Plan to Share IPD: Yes
We plan to share IPD in due course after the study is completed and published.
Supporting Information: Study Protocol, SAP
Time Frame: 36 months after study completion.
Access Criteria: We will attempt to post the data in a public data archive.

REFERENCES:
- [Derived] Goyal M, Ospel JM, Ganesh A, Dowlatshahi D, Volders D, Mohlenbruch MA, Jumaa MA, Nimjee SM, Booth TC, Buck BH, Kennedy J, Shankar JJ, Dorn F, Zhang L, Hametner C, Nardai S, Zafar A, Diprose W, Vatanpour S, Stebner A, Bosshart S, Singh N, Sebastian I, Uchida K, Ryckborst KJ, Fahed R, Hu SX, Vollherbst DF, Zaidi SF, Lee VH, Lynch J, Rempel JL, Teal R, Trivedi A, Bode FJ, Ogungbemi A, Pham M, Orosz P, Abdalkader M, Taschner C, Tarpley J, Poli S, Singh RJ, De Leacy R, Lopez G, Sahlas D, Chen M, Burns P, Schaafsma JD, Marigold R, Reich A, Amole A, Field TS, Swartz RH, Settecase F, Lenzser G, Ortega-Gutierrez S, Asdaghi N, Lobotesis K, Siddiqui AH, Berrouschot J, Mokin M, Ebersole K, Schneider H, Yoo AJ, Mandzia J, Klostranec J, Jadun C, Patankar T, Sauvageau E, Lenthall R, Peeling L, Huynh T, Budzik R, Lee SK, Makalanda L, Levitt MR, Perry RJ, Hlaing T, Jahromi BS, Singh P, Demchuk AM, Hill MD; ESCAPE-MeVO Investigators. Endovascular Treatment of Stroke Due to Medium-Vessel Occlusion. N Engl J Med. 2025 Apr 10;392(14):1385-1395. doi: 10.1056/NEJMoa2411668. Epub 2025 Feb 5. PMID 39908448
- [Derived] Ospel JM, Dowlatshahi D, Demchuk A, Volders D, Mohlenbruch M, Nimjee S, Kennedy J, Buck B, Shankar JJ, Booth TC, Jumaa MA, Fahed R, Ganesh A, Zhang Q, Doram C, Ryckborst KJ, Hill MD, Goyal M; ESCAPE-MeVO investigators. Endovascular treatment to improve outcomes for medium vessel occlusions: The ESCAPE-MeVO trial. Int J Stroke. 2024 Oct;19(9):1064-1070. doi: 10.1177/17474930241262642. Epub 2024 Jun 20. PMID 38845180